CLINICAL TRIAL: NCT04909177
Title: oVRcome Self-guided Virtual Reality for Specific Phobias: A Randomized Controlled Trial
Brief Title: oVRcome Self-guided Virtual Reality for Specific Phobias
Acronym: oVRcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Otago (Other)
Collaborators: oVRcome (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: oVRcome specific phobia
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Specific Phobia
MeSH Terms: conditions — Phobia, Specific | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone application (app) in combination with headset (Experimental): The intervention oVRcome is self-help VRET for specific phobia, that is delivered through a smartphone application (app) in combination with headset that holds the smartphone and uses 360º video. oVRcome includes 6 modules of psychoeducation, relaxation, mindfulness, cognitive techniques, exposure through VR, and a relapse prevention module which are aimed to be completed weekly.
  Interventions: Other: Smartphone application (app) in combination with headset
- Waitlist (No Intervention): Participants in the waitlist condition will be offered the intervention directly after post-test.

INTERVENTIONS:
Other: Smartphone application (app) in combination with headset — The intervention oVRcome is self-help VRET for specific phobia, that is delivered through a smartphone application (app) in combination with headset that holds the smartphone and uses 360º video. oVRcome includes 6 modules of psychoeducation, relaxation, mindfulness, cognitive techniques, exposure through VR, and a relapse prevention module which are aimed to be completed weekly.
  Arms: Smartphone application (app) in combination with headset

SUMMARY:
Specific phobias: fear of flying, heights, spiders, dogs and needles are the extremely common and exposure therapy (ET) is the first line of treatment. Using Virtual Reality (VR), participants will have control in gradual exposure to their fears. oVRcome (https://www.ovrcome.io/ Virtual reality app), is a self-help VRET for specific phobias, that is delivered through a smartphone application (app) in combination with a low cost headset that holds the smartphone and uses 360º video. The investigators hypothesize that oVRcome is effective in reducing specific phobia symptoms.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* are between 18-64 years old
* Have a fear of flying, heights, spiders, dogs, needles and score above 4 on the Brief Standard Self rating scale for phobic patients (Marks, I. Matthews ,A (1979) Behaviour Research and Therapy)
* have access to a smart phone and internet
* willing to participate in the research study and providing informed consent

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* present with symptoms of severe depression or suicidality respectively as measured with the PHQ-9; total score > 19
* have insufficient knowledge of the English language
* are under current treatment for specific phobia or psychotropic medication (unless on stable dosage for the previous 3 months and no changes planned during the study period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Severity Measure for Specific Phobia-Adult American Psychological Association | Week 6
  The Severity Measure for Specific Phobia-Adult is a 10-item self-report measure that assesses the severity of specific phobia in individuals age 18 and older.
  The total score can range from 0 to 40 with higher scores indicating greater severity of specific phobia.

SECONDARY OUTCOMES:
Brief Standard Self rating scale for phobic patients | 6 weeks, 12 weeks, 18 weeks
  The total score can range from 0 to 8 with higher scores indicating greater severity of specific phobia
Clinical Global Impression of Change (CGI-C) | weekly (Weeks 1-6)
  CGI-C scores range from 1 (very much improved) through to 7 (very much worse)
Patient Health Questionnaire - PHQ 9 | 6 weeks, 12 weeks, 18 weeks
  PHQ-9 scores range from 1 through to 27, with higher scores indicating more severe depressive symptoms
Subjective Units of Distress Scale | Week 4, 5 and 6
  Scores range from 1 through to 100 with higher scores indicating higher levels of distress
Modified Gatineau Presence Questionnaire First item | Week 4, 5 and 6
  Scores range from 1 (very realistic) through to 100 (not very realistic)
Fast Motion Sickness Scale (FMS) | Week 4, 5 and 6
  Scores range from zero (no sickness at all) to 20 (frank sickness).
Brief Fear of Negative Evaluation Scale | 6 weeks, 12 weeks, 18 weeks
  Scores range from 1 through to 60 with higher scores indicating higher fear of negative evaluation
Changes in behaviour that may have been previously avoided because of the phobia | Weeks 6 and 12
  Free text response

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Lacey, PhD, Principal Investigator — University of Otago
Locations (1):
- University of Otago, Christchurch, Christchurch, Canterbury, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lacey C, Frampton C, Beaglehole B. oVRcome - Self-guided virtual reality for specific phobias: A randomised controlled trial. Aust N Z J Psychiatry. 2023 May;57(5):736-744. doi: 10.1177/00048674221110779. Epub 2022 Jul 11. PMID 35818296